CLINICAL TRIAL: NCT00071214
Title: A Phase 3, Multicenter, Randomized, Placebo-Controlled, Double-Blinded Study to Evaluate Efficacy of StaphVAX, a Bivalent Staphylococcus Aureus Glycoconjugate Vaccine in Adults on Hemodialysis
Brief Title: Study to Evaluate the Effectiveness of StaphVAX in Adults on Hemodialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nabi Biopharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Nabi-1371
Record Dates: First submitted 2003-10-15; First posted 2003-10-17 (Estimated); Last update posted 2006-07-11 (Estimated); Status verified 2006-07

CONDITIONS: Staphylococcal Infections; Kidney Failure, Chronic
Keywords: Staphylococcal infection; Gram positive bacteria; Staphylococcus; Staphylococcus aureus; Staphylococcus aureus infection
MeSH Terms: conditions — Staphylococcal Infections; Kidney Failure, Chronic

INTERVENTIONS:
Biological: S. aureus Type 5 and 8 Capsular Polysaccharide Conjugate Vaccine

SUMMARY:
Two part study testing the effectiveness and safety of StaphVAX vaccine in chronic hemodialysis patients against infection by Staphylococcus aureus.

DETAILED DESCRIPTION:
Two part clinical trial designed to evaluate the efficacy of StaphVAX in adults on hemodialysis. Part A will evaluate the prevention of bacteremic infections in End Stage Renal Disease (ESRD) patients during the interval between 3 and 35 weeks after a single dose of StaphVAX. Part B of this study is designed to assess immunogenicity of a second [booster] dose of vaccine in patients completing Part A, and the cumulative (Part A + B) efficacy.

ELIGIBILITY:
Eligible subjects must already be receiving chronic hemodialysis treatment from the centers participating in this study. Interested subjects should discuss enrollment with their nephrologist.

Inclusion Criteria:

* Age 18 years or older.
* Diagnosis of chronic end-stage renal disease with maintenance on hemodialysis continuously for at least eight (8) weeks prior to enrollment.
* Hemodialysis access using native vessel fistula or synthetic/heterologous graft (not catheter).
* Expectation of compliance with protocol procedures, and visit schedule.
* Negative serum pregnancy test in females of child-bearing potential (serum -HCG within 7 days prior to each study drug injection).
* Written informed consent.

Exclusion Criteria:

* Known serious S. aureus infection within 3 months of study entry.
* Known recurrent S. aureus infection of the current graft.
* Known active viral or bacterial infection or symptoms/signs consistent with such an infection with the two weeks prior to injection of investigational product. Mild intercurrent viral illness with a temperature of 100.6F or less does not require exclusion, if in the judgement of the investigator this illness will not interfere with the evaluation of the vaccine.
* Known HIV infection (testing not required for protocol).
* Known hypersensitivity or previous anaphylaxis to polysaccharides or polysaccharide-conjugate vaccines or to components of such vaccines.
* Known or suspected abuse of any drugs, prescribed or illicit, in the past year.
* Current use of immunosuppressive or immunomodulatory drugs (including systemic glucocorticoids, chlorambucil, cyclophosphamide, azathioprine, methotrexate, cyclosporine, mycophenolate, human immune globulin in excess of 0.2 g/Kg per month, any monoclonal antibody specific for any human leukocyte subset or cytokine, or any interferon preparation), except low-dose physiologic replacement glucocorticoid therapy (Less than or equal to 10 mg of prednisone or equivalent per day).
* Known malignancy or treatment for malignancy within the past six months, other than basal cell or squamous cell carcinoma of the skin.
* Use of investigational drugs, products, or devices within 30 days prior to vaccine injection.
* Presence of any condition which, in the opinion of the investigator, places the subject at undue risk or potentially jeopardized the quality of the data to be generated.
* Previous administration of StaphVAX

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3600
Dates: Start 2003-09; Study Completion 2005-09

PRIMARY OUTCOMES:
Documented S. aureus invasive infection, weeks 3-35

SECONDARY OUTCOMES:
Documented S. aureus invasive infection in other time periods
Immunogenicity at mulitple time points
Safety
Health economics

CONTACTS AND LOCATIONS:
Overall Officials: Matt Hohenboken, MD, PhD, Study Director — Nabi Biopharmaceuticals

REFERENCES:
- [Derived] Fattom A, Matalon A, Buerkert J, Taylor K, Damaso S, Boutriau D. Efficacy profile of a bivalent Staphylococcus aureus glycoconjugated vaccine in adults on hemodialysis: Phase III randomized study. Hum Vaccin Immunother. 2015;11(3):632-41. doi: 10.4161/hv.34414. PMID 25483694
- [Derived] Li Y, Friedman JY, O'Neal BF, Hohenboken MJ, Griffiths RI, Stryjewski ME, Middleton JP, Schulman KA, Inrig JK, Fowler VG Jr, Reed SD. Outcomes of Staphylococcus aureus infection in hemodialysis-dependent patients. Clin J Am Soc Nephrol. 2009 Feb;4(2):428-34. doi: 10.2215/CJN.03760708. Epub 2008 Dec 31. PMID 19118117